CLINICAL TRIAL: NCT06414954
Title: A Phase 2b, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of 3 Dose Levels of NMD670 Over 21 Days in Adult Patients With AChR/MuSK-Ab+ Myasthenia Gravis
Brief Title: Safety and Efficacy of 3 Dose Levels of NMD670 in Adult Patients With Myasthenia Gravis
Acronym: SYNAPSE-MG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NMD Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMD670-02-0002; 2023-507539-40 (Other: EUCTR)
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis; Myasthenia Gravis, MuSK
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NMD670 high dose (Experimental)
  Interventions: Drug: NMD670
- NMD670 mid dose (Experimental)
  Interventions: Drug: NMD670
- NMD670 low dose (Experimental)
  Interventions: Drug: NMD670
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NMD670 — Tablets taken twice a day for 21 days
  Arms: NMD670 high dose; NMD670 low dose; NMD670 mid dose
Drug: Placebo — Tablets taken twice a day for 21 days
  Arms: Placebo

SUMMARY:
This Phase 2 proof-of-concept, dose range finding study aims to evaluate the safety and efficacy of 3 dose levels of NMD670 vs placebo in adult patients with MG with antibodies against AChR or MuSK, administered twice a day (BID) for 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a male or female being 18 or more, at the time of signing the informed consent
* Diagnosis of MG, MGFA class II, III or IV
* Documented positive AChR or MuSK antibody test.
* Participant must be able to swallow tablets
* Body mass index between 18 and 35 kg/m2, inclusive, at screening, and with a minimum weight of 40 kg
* Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Participant is capable of and has given signed informed consent

Exclusion Criteria:

* Known medical or psychological condition(s) or risk factor that, in the opinion of the Investigator, might interfere with the patient's full participation in the study, pose any additional risk for the patient, or confound the assessment of the patient or outcome of the study
* Participants with other significant clinical and/or laboratory safety findings that may interfere with the conduction or interpretation of the study
* Participants that received treatment with an investigational medical product within 30 days or 5 half-lives of the medication, whichever is longer prior to Day 1
* Participants with history of poor compliance with relevant MG therapy
* Female patients who plan to become pregnant during the study or are currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to day 21 in QMG total score for NMD670 vs placebo | Baseline to day 21
  Scale goes from 0-39 and higher score indicates worse symptomatology

SECONDARY OUTCOMES:
Change from baseline to day 21 in MG-ADL total score for NMD670 vs placebo | Baseline to day 21
  Scale goes from 0-24 and higher score indicates worse symptomatology
Change from baseline to day 21 in MGC total score for NMD670 vs placebo | Baseline to day 21
  Scale goes from 0-50 and higher score indicate worse symptomatology
Change from baseline to day 21 in MG-QOL15r for NMD670 vs placebo | Baseline to day 21
  Scale goes from 0-30 and higher score indicate worse quality of life
Change from baseline to day 21 in Neuro-QoL Fatigue Short Form | Baseline to day 21
  Scale goes from 8-40 and higher score indicate worse symptomalogy
Incidence of treatment emergent adverse event | Over 21 days of dosing
  Summarised per treatment
Incidence of serious treatment emergent adverse events | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on physical examinations | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on safety laboratory parameters | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant vital signs abnormalities | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant ECG abnormalities | Over 21 days of dosing
  Summarised per treatment
Incidence of Suicidal Ideation or Suicidal Behavior | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on opthalmological examinations | From screening (day -28 to day -1) until follow up (day 28)
  Summarised per treatment

CONTACTS AND LOCATIONS:
Locations (39):
- United States (11):
  - Profound Research LLC, Carlsbad, California
  - University of California Irvine Medical Center, Irvine, California
  - University of Colorado Neuromuscular Division, Aurora, Colorado
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Neuromuscular Research Division | University of South Florida, Tampa, Florida
  - Augusta University, Neuroscience Center, Augusta, Georgia
  - NextGen Precision Health, Columbia, Missouri
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Oregon, Portland, Oregon
  - Semmes Murphey Clinic, Memphis, Tennessee
- UZ Leuven, Leuven, Belgium
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet University of Copenhagen, Copenhagen
- France (5):
  - Centre de référence des maladies neuromusculaires AOC-CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Centre de Référence des Maladies Neuromusculaires et de la SLA, Marseille
  - Centre Hospitalier Universitaire de Nantes - Hôtel Dieu Centre de Référence des Maladies Neuromusculaires Rares -, Nantes
  - CHU de Nice, Nice
  - Unité de Recherche Clinique NeuroSciences, Nice
- Georgia (3):
  - JSC Curatio, Tbilisi
  - LTD David Tatishvili Health Center, Tbilisi
  - Ltd New Hospitals, Tbilisi
- Italy (8):
  - ASST Papa Giovanni XXIII (Azienda Ospedaliera Papa Giovanni XXIII), Bergamo
  - IRCCS Istituo delle Scienze neurologiche di Bologna, UOC Clinica neurologica Ospedale, Bologna
  - IRCCS Ospedale Policlinico San Martino, Genova
  - IRCCS Fondazione Istituto Neurologico Carlo Besta, Dipartimento di Ricerca e Sviluppo clinico, Milan
  - DIMER, IRCCS, Ospedale San Raffaele, Milan
  - Centro Sclerosi Multipla Napoli - AOU Vanvitelli, Napoli
  - AOU Pisana, Pisa
  - Azienda Ospedaliera Sant'Andrea - Universita di Roma La Sapienza, Roma
- Leiden Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- Poland (5):
  - Neurologia Śląska Centrum Medyczne, Katowice
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie sp.z o.o, Krakow
  - Centrum Medyczne Hope Clinic, Lublin
  - Galen Clinic, Lublin
  - Centrum Medyczne Neuro Protect, Warsaw
- Serbia (2):
  - University Clinical Center of Serbia, Neurology Clinic, Belgrade
  - University Clinical Center Nis, Neurology Clinic, Niš
- Hospìtal Universitari Vall d'Hebrón, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No